CLINICAL TRIAL: NCT02837861
Title: Early Metabolomic Support Study
Brief Title: Early and Adequate Protein Feeding Post-Traumatic Injury
Acronym: EMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-34322; 1R21DK108145-01A1 (NIH)
Record Dates: First submitted 2016-06-29; First posted 2016-07-20 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Protein Feeding in Post-traumatic Injury Patients
Keywords: Metabolic Support; Nutritional Support; Neuro-endocrine Event; Enteral feedings; Parenteral feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Routine Nutritional Support plus supplemental IV amino acids, to begin within 24h of injury. (Target approximately 1.5-2g protein/kg/day)
  Interventions: Drug: Routine Nutritional Support plus supplemental IV amino acids
- Control Group (Active Comparator): Routine Nutritional Support (i.e. enteral nutrition as tolerated, to begin as early as medically feasible)
  Interventions: Other: Routine Nutritional Support

INTERVENTIONS:
Drug: Routine Nutritional Support plus supplemental IV amino acids — Enteral nutrition as tolerated Plus supplemental IV AA infusion to meet the target of approximately 1.5-2.0gm protein/kg/day total starting within 24 hours of injury for 5 days.
  Other Names: Plenamine
  Arms: Experimental Group
Other: Routine Nutritional Support — Enteral nutrition as tolerated.
  Arms: Control Group

SUMMARY:
A randomized, parallel-group, pilot study comparing the effect of the early addition of intravenous protein to enteral feeding as tolerated versus enteral feedings as tolerated alone immediately post traumatic injury.

Primary: To determine that early and adequate nutritional support will improve protein economy in the first week post -injury as measured by nitrogen balance. We hypothesize that an improvement in nitrogen balance with early maximized protein intake will support the production of acute phase proteins, major antioxidants and the inflammatory response.

Secondary: Through the use of mass spectrometry (MS) and nuclear magnetic resonance (NMR) technologies we will determine that our plan for early and adequate nutritional support with adequate protein from day one post injury will alter the metabolomics profile when compared to routine nutritional support.

Tertiary: For Specific Aim 3 we will measure several pro- and anti-inflammatory cytokines and soluble proteins.

DETAILED DESCRIPTION:
* Subjects admitted to the trauma service and cared for in the SICU will be screened for participation in this study.
* If subjects meet eligibility criteria, they will be enrolled and randomized 1:1 to enteral nutrition alone or enteral nutrition plus Amino Acid (AA) infusions.
* Nutritional assessment will be completed.
* Various procedures/assessments will take place over the course of the trial.
* Subjects will be followed for 28 days or until discharged or disposition of status.

Potential subjects deemed eligible will be randomized by the REDCap Randomization Module and begin study interventions within the first 24 hours of admission to the Surgical Intensive Care Unit (SICU).

Subjects enrolled into the Control Arm will receive routine nutritional support (RNS). RNS for the purpose of this study is defined as:

* Nutrition delivered via the enteral route of administration;
* Enteral caloric goal of 60-80% of energy requirements;
* Enteral feedings to be initiated as soon as medically feasible;
* Full parenteral nutrition to be initiated on Day 7 if enteral nutrition has not been started. Subjects will complete the study after Day 5 and will continue with nutritional support as clinically indicated.

Subjects enrolled into the Experimental Arm will receive RNS plus supplemental intravenous amino acids (RNS+IVAA). RNS+IVAA for the purpose of this study is defined as:

* Nutrition delivered via the enteral route of administration;
* Enteral caloric goal of 60-80% of energy requirements;
* Enteral feedings to be initiated as soon as medically feasible;
* Full parenteral nutrition to be initiated on Day 7 if enteral nutrition has not been started.
* Supplemental intravenous amino acids to begin within 24 hours of admission to the Surgical Intensive Care Unit (SICU);
* Amino acids to supplement enteral protein for total protein intake of approximately 1.5-2g/kg/day. Subjects will complete the study after Day 5 and will continue with nutritional support as clinically indicated.

Allocation of Treatment and Randomization Procedures 40 subjects will be recruited into the study and will be randomized in a 1:1 ratio. This will take place in lots of 10; permitting evaluation of data after every ten subjects. Potential subjects deemed eligible will be randomized in a blinded fashion by the REDCap Randomization Module to receive either routine nutritional support , enteral feedings as soon as medically feasible supplemented with intravenous amino acids " or routine nutritional support enteral feedings as soon as medically feasible. Randomization treatment assignment list will be created by our statistician; taking into consideration drop outs and replacements.

ELIGIBILITY:
Inclusion Criteria:

* Trauma Patient /Male or female, any race/ethnicity
* Expected to survive 72 hours
* Admitted to the SICU
* Expected to remain in the hospital for at least 7 days
* Candidates for enteral nutrition post-injury

Exclusion Criteria:

* BMI less than 18 mg/m2 or greater than 35 mg/m2
* Immunosuppressive disorders (i.e. Prednisone >20mg daily; Organ Transplant Recipient with active immunosuppression treatments, diagnosis of HIV/AIDS).
* Type I or Type II Diabetes
* Pregnancy
* Pre-existing renal dysfunction (creatinine >2.5mg/dL).
* Clear contraindication for enteral nutrition immediately post injury
* Severe liver dysfunction (Total Bilirubin > 3.0mg%)
* Non-English speaking patients
* Known allergies to any of the study drug's components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Nitrogen balance and Catabolic Index | 8 days
  We will use the urine specimen collections to measure nitrogen balance and catabolic index, both of which assess the level of physiologic stress. A catabolic Index less than zero represents no significant stress, an index greater than or equal to zero and less than or equal to 5 represents moderate stress, and an index greater than 5 represents severe stress. Twenty-four hour urine collections will be done for measurement of urine urea nitrogen to estimate nitrogen balance on day 1 and day 5 or 6 or 7 of the study. This will allow us to compare degree of catabolism and nitrogen efficiency between groups as well as between the two time points (Day 1 and Day 5 or 6 or 7). We hypothesize the early and adequate protein feeding group, although receiving fewer overall calories than subjects' total requirements, will have less negative nitrogen balance than the control group.

SECONDARY OUTCOMES:
Metabolomics Profiles | 8 days
  Through the use of mass spectrometry (MS) and nuclear magnetic resonance (NMR) technologies we will determine whether our plan for early and adequate nutritional support with adequate protein from day one post injury will alter the metabolomics profile when compared to routine nutritional support. We expect:
  1. An improvement in protein (specifically branched chain amino acid) utilization with reduced 3-methylhistidine production and decreased proteolysis from peripheral stores;
  2. Improved redox potential as measured by products of oxidation: primarily glutathione precursors and metabolites and products of lipid peroxidation;
  3. Improvement in the lipid milieu seen post injury to reflect expected inflammatory response and not reflect the metabolomics profile observed with developing MODS (i.e. increased glycerol heads of phospholipids as opposed to increased fatty acyl chain, creatinine and lactate).

OTHER OUTCOMES:
Inflammatory Biomarkers | 8 days
  Early and adequate protein support will modify the levels of select pro and anti-inflammatory cytokines levels as compared to standard nutritional care. We anticipate decreased levels of the stress response mediators such as cortisol, Tumor Necrosis Factor (TNF), Interleukin-6 (IL-8)and Interleukin-8 (IL-8). These inflammatory markers are also key regulators of the breakdown of muscle during the acute stress response and their down-regulation would also serve to protect lean muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Burke, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
A Data and Safety Monitoring Safety plan has been created per Boston University Medical Campus (BUMC) guidelines. The Principal Investigator at Boston Medical Center (BMC) or Boston University Medical Campus will report all adverse events and Unanticipated Problems to the Institutional Review Board (IRB) in compliance with IRB policy, Federal/State regulations, and sponsor requirements.

REFERENCES:
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Hill AA, Plank LD, Finn PJ, Whalley GA, Sharpe N, Clark MA, Hill GL. Massive nitrogen loss in critical surgical illness: effect on cardiac mass and function. Ann Surg. 1997 Aug;226(2):191-7. doi: 10.1097/00000658-199708000-00011. PMID 9296513
- [Background] Sandstrom R, Drott C, Hyltander A, Arfvidsson B, Schersten T, Wickstrom I, Lundholm K. The effect of postoperative intravenous feeding (TPN) on outcome following major surgery evaluated in a randomized study. Ann Surg. 1993 Feb;217(2):185-95. doi: 10.1097/00000658-199302000-00013. PMID 8439216